CLINICAL TRIAL: NCT04743128
Title: Impact of Exercise on Expression of Hsp70 in Individuals at Risk of Peripheral Arterial Disease. A Randomised Trial
Brief Title: Exercise on Expression of Heat Shock Protein 70 in Arterial Risk
Acronym: HSP70
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Popular Autónoma del Estado de Puebla (Other)
Responsible Party: Principal Investigator, Clara Luz Pérez Quiroga, MSc, Universidad Popular Autónoma del Estado de Puebla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSP 70 CLPQ
Record Dates: First submitted 2021-01-27; First posted 2021-02-08 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Aerobic Exercise; HSP70
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group received written recommendations to exercise three times per week, for a period of 12 weeks but they did not attend the training sessions.
- Exercise group (Experimental): The experimental group started an exercise program to achieve 65% to 80% of the maximum heart rate by using a pulsometer that measured the heart rate in order to get to the moderate intensity activity goal. The exercise session was 60 minutes long, three times per week, completing 180 minutes per week of moderate intensity exercise, for 12 weeks in total.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The experimental group started an exercise program to achieve 65% to 80% of the maximum heart rate by using a pulsometer that measured the heart rate in order to get to the moderate intensity activity goal. The exercise session was 60 minutes long, three times per week, completing 180 minutes per week of moderate intensity exercise, for 12 weeks in total.
  Arms: Exercise group

SUMMARY:
Introduction: Atherosclerotic Peripheral Arterial Disease (PAD) is the leading cause of mortality in the western world. To maintain homeostasis of the vessel wall, vascular cells produce a high level of heat shock proteins (HSP), among which is Hsp70, to stimulate innate immunity and face stress.

Methods: This is a clinical trial where 260 individuals were evaluated by a screening test employing the Ankle-Arm Index (ABI), 220 of them were not within risk value (0.91 to 0.99 mmHg). In the clinical trial, 32 individuals were included. A control group and an experimental group were formed. Aerobic exercise intervention was performed for 12 weeks. The level of Hsp70 was evaluated, physical and clinical measurements were applied at the beginning and at the end of the trial.

DETAILED DESCRIPTION:
The objective of the study is to determine the level of serum expression of the HSP70 protein in individuals at risk of atherosclerotic peripheral arterial disease, after an intervention of moderate exercise.

Atherosclerotic Peripheral Arterial Disease (PAD) is a systemic disease that causes obstruction of arterial blood flow and is a significant cause of morbidity and mortality worldwide 1.

Patients with PAD have a three times greater risk of myocardial infarction, stroke and death than those without the disease. However, more than 50% of patients are asymptomatic; so the disease remains underdiagnosed. 2 It is estimated that 202 million people in the world are affected with PAD, 45 million of them die from coronary or cerebrovascular disease in a range of ten years. The current prevalence of PAD in Mexico is 10% of the general population.3 The disease is strongly related to modifiable risk factors (blood pressure, sedentary lifestyle, baseline glycemia, cholesterol, and obesity) and unhealthy lifestyle (tobacco, physical inactivity, food and psychosocial stress), which increases the risk of acquiring the disease up to 17.2 times 4, 5, 6 Increased membrane permeability leads to the accumulation and modification of proteins, lipids and lipoproteins in the endothelium. The accumulation of pro-inflammatory molecules such as chemo-tactical monocyte protein 1 (MCP-1), intracellular adhesion molecules (ICAM-1), vascular cell adhesion (VCAM-1) and higher nitro-tyrosine content are also generated. 7 Macrophages are active in response to the spread of the inflammatory response and bind to low-density lipoprotein (LDL) receptors that had internalized.

Macrophages secrete pro-inflammatory cytokines resulting in the recruitment and activation of additional immune cells at the site of the lesion, amplifying the immune response and promoting the development of complex and advanced plaques that become mature atherosclerotic plaques.8 The Ankle Arm Index (ABI) is the non-invasive gold standard accepted for both the diagnosis and evaluation of the severity of this disease. The cut-off point for the diagnosis of PAD is an ABI of less than 0.90 at rest, regardless of the Framingham Risk Score, being 95% sensitive in the detection of PAD. 9, 10 To maintain homeostasis on the vessel wall, vascular cells produce a high level of heat shock proteins (HSP) 11. These types of stress proteins are cytoprotective agents that promote cell survival during stressors. 12 The reduction of HSP intracellular expression is also related to PAD, cardiovascular diseases and metabolic syndrome, where they are greatly diminished. 10 HSP are normally intracellular proteins, but when released at an extracellular level, they exert an immune response.13 The most thermo-sensitive and highly inducible HSP belongs to the 70 kilodalton (kDa) family, as established by Mizzen et al., In 1998 (figure 1). It is believed that extracellular Hsp70 (eHsp70) stimulates innate immunity and acts as a danger signal. Serum Hsp70 has been detected in the peripheral circulation of apparently healthy individuals and increases in response to different stressors, including exercise. 12, 14

Figure 1. Schematic representation of the molecular structure of HSP70. Adapted from Carrasco L. et al. 15 Exercise increases HSP levels primarily through reactive oxygen species (ROS), elevated temperature, hormones, calcium fluxes or mechanical tissue deformation.16 It has been shown that the concentration of Hsp70 increases after performing both acute and long-term exercises, reaching levels that remain high, but once its protective action decreases both at intra and extra-cellular levels.17 Exercise exerts beneficial effects against atherosclerosis by increasing circulating endostatin, which inhibits the development of atherosclerotic plaque by blocking angiogenesis in plaque tissue.18 Isotonic contractions of the type of resistance exercise (aerobic) tend to lead to increases in Hsp70 levels, as opposed to eccentric exercise. With repetitive exercise, an induced increase in this protein is maintained, while the initial response of other HSPs to exercise decreases as training progresses.16 Regular exercise initiates long-term processes of adaptation of muscle metabolism, cardiovascular system and immuno-modulatory effects that are largely considered beneficial; There is evidence that during exercise, Hsp70 is released into human circulation in association with exosomes, specifically with aerobic exercise.19, 20 It has been shown that Hsp70 directly inhibits inflammatory processes through the suppression of oxidative stress, directly reduces apoptosis, hyperplasia, as well as decreasing the expression of adhesion molecules that lead to leukocyte extravasation and the manifestation of inflammatory cytokines.16 Higher serum levels of Hsp70 are associated with reduced thickening of the atherosclerotic intima and a lower risk of coronary artery disease.21

ELIGIBILITY:
Individuals who attended the internal medicine service of the "Instituto de Seguridad y Servicios Sociales para los Trabajadores del Estado de Puebla" (ISSSTEP) Hospital were invited to participate voluntarily, from February to September of 2019. In order to detect people at risk of PAD, the measurement of the ABI was done. The measure was taken after 10 minutes of resting. The measure was taken in the four extremities to obtain systolic BP of the posterior tibial artery and brachial artery. The cut point to enter the study was between 0.91 and 0.99 mmHg. The informed consent was signed by all the individuals.

Inclusion criteria

* ABI cut point from 0.91 to 0.99
* Age, from 40 to 75 years old
* Both genders

Exclusion criteria

* Unable to perform Bruce's stress test
* Presence of fractures or sprains in the last 3 months
* Diagnosis of diabetes, heart disease, angina pectoris or heart attack

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Impact of exercise on expression of Hsp70 in individuals at risk of peripheral arterial disease | 12 weeks
  This is a clinical trial where 260 individuals were evaluated by a screening test employing the Ankle-Arm Index (ABI). A number of 220 individuals were not within risk value (0.91 to 0.99 mmHg). In the clinical trial, 32 individuals were included. A control group and an experimental group were formed. Aerobic exercise intervention was performed by the experimental group. The level of Hsp70 was evaluated, physical and clinical measurements were applied at the beginning and at the end of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Luz Pérez Quiroga, MCs, Principal Investigator — Universidad Popular Autónoma del Estado de Puebla
Locations (1):
- UPAEP, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT04743128/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT04743128/SAP_001.pdf
  • Informed Consent Form (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT04743128/ICF_000.pdf